CLINICAL TRIAL: NCT03849937
Title: Changing Talk Online (CHATO): A Pragmatic Trial to Reduce Behavioral Symptoms in Dementia Care
Brief Title: Changing Talk Online (CHATO) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1R61AG061881-01 (NIH)
Record Dates: First submitted 2019-01-22; First posted 2019-02-21 (Actual); Results first posted 2021-08-19 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-08

CONDITIONS: Staff Attitude; Dementia
Keywords: Behavioral and Psychological Symptoms of Dementia; Psychotropic Medication; Elderspeak; Staff Training; Staff Communication; Nonpharmacological treatment for Dementia
MeSH Terms: conditions — Dementia; Behavior

STUDY DESIGN:
Intervention Model Description: The research design is a randomized clinical trial. An initial nursing home will be used to test feasibility. Six nursing homes will be randomly assigned to intervention or wait-list control groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Three nursing homes will receive the training and three control nursing homes will complete assessments, but not receive the training.
  Interventions: Behavioral: Changing Talk Online (CHATO)
- Waitlist Control (Active Comparator): After the intervention group takes the training, the waitlist control group will crossover and take the training.
  Interventions: Behavioral: Changing Talk Online (CHATO)

INTERVENTIONS:
Behavioral: Changing Talk Online (CHATO) — Three, one-hour online training modules highlighting barriers and ineffective communication behaviors with older adults while teaching and modeling alternative, effective communication strategies.

SUMMARY:
Objectives AIM 1. Establish acceptability and preliminary efficacy of online CHATO modules through pilot testing with NH staff.

AIM 2. Develop and pilot test the data collection tool with consultant and advisory panel input. Interviews of NH administrators and staff who participate in the pilot testing of CHATO and a process evaluation will be used to identify and develop supports for implementation and sustainability in preparation for future CHATO testing.

Design and Outcomes The R61 will prepare for the R01 pragmatic trial by establishing feasibility of online modules and preliminary efficacy of CHATO with NH staff. The research design is a randomized clinical trial. One NH will provide initial feasibility testing. Any modifications to the modules will be made. Then six nursing homes (estimated N=150 staff) will be randomly assigned to intervention or wait-list control groups. The primary outcome will be knowledge gain for staff completing CHATO training. Additional outcomes include resident quality measures related to behavioral and psychological symptoms of dementia (BPSD) on both resident and facility levels and facility level data related to inappropriate use of psychotropic medications to control BPSD. Implementation strategies will be assessed by survey and leadership interviews completed by an external evaluator.

Interventions and Duration Changing Talk Online (CHATO) training is a course is to increase awareness of the importance of effective communication with older adults and to use evidence-based person-centered communication during interactions with older adults in nursing homes and other health care settings. The total program is approximately 3 hours, split into 3 modules. Each module is approximately an hour, depending on the individual user. Each NH will work with the research team for three months to plan, implement, and collect data.

Sample Size and Population This course is designed for staff in nursing homes, independent and assisted living, and health care settings in the community that include registered nurses, nursing assistants, nursing home dieticians, direct care professionals, other administrations and support employees. All the employees at all seven nursing homes will be asked to participate. Assignment of NHs to intervention and wait-list control groups will be at random. A sample of 150 training participants are estimated.

DETAILED DESCRIPTION:
Background on Condition, Disease, or Other Primary Study Focus: The population afflicted with Alzheimer's disease and other dementias will expand from 5 to 16 million by 2050, increasing dementia care costs from $259 billion to $1.1 trillion. Of today's 1.4 million nursing home (NH) residents, 61% have moderate to severe dementia, and up to 90% of them exhibit behavioral and psychological symptoms of dementia (BPSD) such as physical and verbal aggression, agitation, and wandering. These behaviors are associated with depression as well as reduced quality of life and lower survival rates in persons with dementia (PWD). BPSD also stress family caregivers and precipitate NH placement. In the NH, BPSD increase time to provide care, and NH staff, primarily Certified Nursing Assistants (CNAs) who provide most direct care, report that BPSD represent the most stressful aspect of their job. Considering additional costs for CNA burnout and turnover, It is estimated that BPSD increase costs of dementia care by 25 to 35%. With national NH rates for a semi-private room of $82,200 per year, reducing BPSD may save up to $20,000 per resident annually.

As cognitive and communication abilities decline due to dementia, NH residents become unable to convey care preferences and needs and staff communication becomes infantilizing, impersonal, and task-oriented resulting in BPSD. As verified in the investigator's past research using behavioral coding and sequential analyses of video-recorded care, staff elderspeak (communication that sounds like baby talk) is linked to resident resistiveness to care (RTC), a subset of BPSD that disrupt nursing care. NH residents were more than twice as likely to be resistive to care when staff used elderspeak compared to normal communication. Thus, improving communication has great potential as a nonpharmacological intervention to reduce BPSD in NH care.

Study Rationale: The Communication Predicament of Aging theory establishes the link between elderspeak and BPSD. Elderspeak derives from stereotypical views of older adults as less competent than younger persons. When younger people talk with older adults, they modify their speech by simplifying, clarifying, and altering the underlying affective quality of messages. The resulting implicit message of incompetence begins a negative feedback loop for older persons, who react with depression, withdrawal, and dependency. Elderspeak is especially threatening to self-concept and personhood, critical to the wellbeing of PWD who are likely to respond with BPSD. The Need-driven Dementia-compromised Behavior model recognizes BPSD as the expression of unmet needs of PWD. Communication, that staff can modify to prevent BPSD, is an essential constant part of the environment connecting PWD to others and affirming their self-concept.

Psychotropic medications are often used inappropriately to control BPSD in NH residents with dementia. Alarmingly high rates persist, despite negative outcomes, an FDA black box warning of increased mortality for older adults with dementia, and a recent Centers for Medicare and Medicaid Services (CMS) mandate to reduce off-label prescribing of antipsychotics. CMS and the National Partnership to Improve Dementia Care target reductions in psychotropic drug use as top priority. Despite reductions in antipsychotic rates (one type of psychotropic medication) ranging from 3 to 12% from 2011-2016, up to 20% of NH residents received inappropriate antipsychotic medication in 2017. Research demonstrates that educating direct care providers in behavioral interventions to control BPSD also reduces psychotropic drug use (antipsychotics, hypnotics, antidepressants, antianxiety, sedative, anticonvulsant and mood stabilizers), although evidence is limited by lack of rigorous clinical trials that also evaluate approaches that influence intervention effects.

The recently completed R01 clinical trial that tested Changing Talk (CHAT) communication training (NR011455) provides preliminary data for this CHATO pilot. CHAT decreased staff elderspeak that reduced resident RTC and increased staff awareness of elderspeak's negative effects. CHAT NHs also saw a significant reduction in psychotropic medication use after the training versus averaged state rates. Despite the success of CHAT in reducing elderspeak and RTC, investigators found challenges to educating NH staff that limited participation in CHAT including turnover, absenteeism, heavy workloads, and personal conflicts. Each CHAT session was held multiple days and times. Still, as few as 44% of staff in one NH completed at least two of the three sessions, although this rate is higher than that noted for other NH staff training programs. Although successful in reducing RTC, the classroom format limits staff access and participation and feasibility for widespread dissemination. Creative, efficient approaches are needed to overcome NH staff education barriers. An online web conference training with multiple NHs as an alternative format was first evaluated for increasing access and dissemination. However, engagement of individual staff was limited with this approach. To facilitate dissemination, online CHAT modules (CHATO) were developed to provide the same CHAT content with asynchronous and independent access for busy NH staff.

The PI worked with an instructional designer, item writer, and media team to transition CHAT content, including 20 video clips of NH staff-resident interactions, to the online CHATO modules. Scripts from the original CHAT were narrated to maintain content, integrating adult learning theories and principles for online learning, and eliminating a need for advanced literacy skills. Interactive scenario and game-based activities engage staff. For example, participants watch a video clip, select problem communication in the transcript, type their improved communication, and compare it to suggested corrections. Moderated online discussions are included in the modules that are supported on Training-Source.org, a free and publicly available learning portal. IT functionality and content equivalency of the newly developed CHATO online modules was demonstrated by a convenient university-affiliated sample of nurses, CNAs, and students with NH experience. Although the group testing CHATO may not represent all NH staff, findings confirm that CHATO is feasible and comparable in content and effects.

While CHAT effectively reduced RTC, the in-person classroom format required an onsite interventionist, which limits accessibility and feasibility for dissemination. A pilot test of acceptability and preliminary efficacy of online CHATO modules is the next logical step. The pilot will prepare for a pragmatic clinical trial that will test the effects of improved staff communication (from CHATO) on resident BPSD and effects on psychotropic medication use. This research will address the gap in rigorous trials testing nonpharmacological interventions to decrease BPSD that also identify strategies to improve intervention dissemination. The goal is to increase access to CHATO training, as a tool to reduce BPSD and inappropriate psychotropic medication use to improve dementia care.

STUDY DESIGN

The R61 will prepare for the R01 pragmatic trial by establishing feasibility of online modules and preliminary efficacy of CHATO with NH staff. The research design is a randomized clinical trial. One NH will provide initial feasibility testing. Any modifications to the modules will be made. Then 6 nursing homes (estimated N=150 staff) will be randomly assigned to intervention or wait-list control groups. The primary outcome will be knowledge gain for staff completing CHATO training. Additional outcomes include resident quality measures related to behavioral and psychological symptoms of dementia (BPSD) on both resident and facility levels and facility level data related to inappropriate use of psychotropic medications to control BPSD.

Staff Knowledge Gain. At time 1, nursing home staff in both groups will complete baseline pre-tests of knowledge and rating of communication. The immediate intervention group will then complete the online CHATO modules within a one-month period. This includes assessments of post-test knowledge, communication rating, program evaluation, and diffusion of innovation surveys at Time 2. Also, at Time 2, the wait-list control group will repeat the pre-tests of knowledge and communication rating and will then complete the CHATO online module training over a one-month period, followed by Time 3 collection of post-test knowledge, communication rating, program evaluation, and diffusion of innovation surveys. Knowledge gain and communication rating data will be compared between the intervention and wait-list control groups and within nursing homes before and after the CHATO training. The immediate and wait-list groups will be compared at baseline to identify important covariates for analyses of changes in outcomes. Changes in knowledge from Time 1 (baseline) to Time 2 will be compared between immediate and wait-list groups using model estimates obtained with a linear mixed model (LMM) approach to account for repeated measures and clustering within nursing homes. Next, pre- to post-training changes in knowledge will be combined for immediate and wait-list groups and also tested using LMM approach.

Resident Quality Measure Outcomes. In addition, nursing homes in both groups will provide monthly summary reports for behavioral symptom occurrence for the facility (in aggregate as well as for individual residents [deidentified]). A nursing home aggregate antipsychotic medication use report will also be collected and analyzed. The BPSD and medication reports will be provided for the one-month period before baseline data collection and for each month thereafter until the post-training assessment of the wait-listed nursing homes is completed (a total of seven months for both groups). Resident outcomes data will be compared between the intervention and wait-list control groups and within nursing homes before and after the CHATO training. Initially, seven months of data will be plotted to examine changes in nursing homes and resident outcomes. Pre- to post-training differences will be compared between immediate and wait-listed groups with a LMM approach.

Implementation Strategies and Process Evaluation. An Implementation Toolkit for NHs and a CHATO Training Manual have been created to provide support and implementation suggestions to pilot nursing homes. Several consultants provided feedback and additional resources to be included in these materials. Each NH will be given a three-month period to complete the CHATO training. One month for orientation, team development, and planning, one month to complete the three-week training, and one month for staff recognition and follow up. The CHATO Research Team will meet with the NH leadership at the beginning and end of this three-month period, manage CHATO training virtual discussion board, and provide technical assistance as necessary. The process evaluation includes an online implementation survey which identifies the strategies NHs used to implement the training and includes the Artifacts of Culture survey. The survey uses the Diffusion of Innovation framework and mirrors the Implementation Toolkit. Additional process evaluation activities include: Leadership phone interviews completed by the consultants and external evaluators at LeadingAge and open-ended questions asked of direct care staff in the CHATO virtual discussion.

ELIGIBILITY:
Inclusion Criteria

* Nursing Homes that serve people with dementia.
* Nursing Homes that have internet available for staff to complete the CHATO training.
* Nursing Homes that are willing to complete leadership interviews and surveys.
* CNAs and nurses who are permanent employees and who provide direct care at least 8 hours weekly will be invited to complete the CHATO training, available by URL link.
* Other personnel, such as housekeeping, dietary, and administrators may also participate. Participation by as many staff as possible is desired to achieve facility-wide communication change.
* Aggregate, deidentified data for residents with Alzheimer's disease or non-Alzheimer's dementia documented on the MDS Active Diagnoses list.

Exclusion Criteria

* Assisted Living facilities or other types of facilities are excluded due to lack of MDS data as well as NHs that previously participated in the CHAT study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Iowa School of Nursing, Iowa City, Iowa
  - University of Kansas School of Nursing, Kansas City, Kansas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Williams KN, Coleman CK, Perkhounkova Y, Beachy T, Hein M, Shaw CA, Berkley A. Moving Online: A Pilot Clinical Trial of the Changing Talk Online Communication Education for Nursing Home Staff. Gerontologist. 2021 Nov 15;61(8):1338-1345. doi: 10.1093/geront/gnaa210. PMID 33346349

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Staff participants at three nursing homes will receive the training and three control nursing homes will complete assessments, but not receive the training.
  Changing Talk Online (CHATO): Three, one-hour online training modules highlighting barriers and ineffective communication behaviors with older adults while teaching and modeling alternative, effective communication strategies.
- Waitlist Control: After the intervention group takes the training, the waitlist control group of staff participants will crossover and take the training.
  Changing Talk Online (CHATO): Three, one-hour online training modules highlighting barriers and ineffective communication behaviors with older adults while teaching and modeling alternative, effective communication strategies.
Period: Overall Study
Arm/Group | Intervention | Waitlist Control
Started | 147 | 72
Completed | 94 | 35
Not Completed | 53 | 37

BASELINE CHARACTERISTICS:
Groups:
- All Direct Care Staff: All staff were encouraged to take the training with a goal of changing the communication culture in each NH. Results are reported for direct care staff, defined as individuals who have daily communication with residents.
Arm/Group | All Direct Care Staff
Number analyzed (Participants) | 219
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 219
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One missing
  Participants
    number analyzed (Participants) | 218
    Female | 203
    Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 153
  Unknown or Not Reported | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 175
  More than one race | 0
  Unknown or Not Reported | 37
Region of Enrollment [Number; unit: participants]
  United States | 219

OUTCOME MEASURES:

1. Primary Outcome: Knowledge Gain Scores for CHATO Training Participants
Description: CHATO Knowledge Test was given to participants pre training and post training. Scoring: 13 items scored incorrect (0) or correct (1). Test score was calculated as the percentage of correct answers (0-100%). The mean percentage was used for each group in the the analysis. Two forms (Forms A and B) measures knowledge gained from training.
Time Frame: Baseline, 1 month, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 94 | 35
score on a scale
  Baseline | 63.0 (17.6) | 58.7 (20.5)
  1 month | 83.8 (13.4) | 63.0 (17.6)
  3 months | NA (NA) — The intervention group completed the training between baseline and 1 month. There is a 3 week washout between baseline and 1 month scores for the waitlist control. The waitlist control crosses over to take the training between 1 month and 3 months. The intervention Group was not evaluated at the three month time point. | 86.8 (13.8)
Statistical Analysis 1: Comparison: Intervention; Test type: Superiority; p < .001, t-test, 2 sided
Statistical Analysis 2: Comparison: Waitlist Control; Test type: Superiority; p = .091, t-test, 2 sided — Time 1 to Time 2
Statistical Analysis 3: Comparison: Waitlist Control; Test type: Superiority; p < .001, t-test, 2 sided — Time 2 to Time 3

2. Primary Outcome: Communication Rating Scores for CHATO Training Participants
Description: Participant watches a video and answers questions testing their ability to visually and audibly identify effective vs ineffective communication strategies and recognize elderspeak vs. person-centered care. Effective rating: mean score for one item scored 1 = Ineffective to 5 = Effective; lower score indicates improvement. Appropriate rating: mean score for one item scored 1 = Inappropriate to 5 = Appropriate; lower score indicates improvement. Recognizes elderspeak subscale: mean score for 6-items scored yes (1) or no (0); higher score indicates improvement. Recognizes person-centered communication subscale: mean score for 3-items scored yes (1) or no (0); lower score indicates improvement.
Time Frame: Baseline (pre-training), 1 month (post-training)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Direct Care Staff - Pre Training: Pre Training results are reported for direct care staff, defined as individuals who have daily communication with residents.
- All Direct Care Staff - Post Training: Post Training results are reported for direct care staff, defined as individuals who have daily communication with residents.
Arm/Group | All Direct Care Staff - Pre Training | All Direct Care Staff - Post Training
Number analyzed (Participants) | 102 | 102
score on a scale
  Effective Communication | 2.7 (1.2) | 2.1 (1.1)
  Appropriate Communication | 3.1 (1.2) | 2.2 (1.1)
  Recognizes Elderspeak | 0.6 (0.2) | 0.7 (0.3)
  Recognizes person-centered communication | 0.5 (0.4) | 0.3 (0.4)
Statistical Analysis 1: Comparison: All Direct Care Staff - Pre Training vs All Direct Care Staff - Post Training; Effective Communication; Test type: Superiority; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: All Direct Care Staff - Pre Training vs All Direct Care Staff - Post Training; Appropriate Communication; Test type: Superiority; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: All Direct Care Staff - Pre Training vs All Direct Care Staff - Post Training; Recognizes elderspeak; Test type: Superiority; p < .001, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: All Direct Care Staff - Pre Training vs All Direct Care Staff - Post Training; Recognizes person-centered communication; Test type: Superiority; p < .001, Wilcoxon (Mann-Whitney)

3. Primary Outcome: BPSD Reports for the One-month Period Before Baseline Data Collection and One Month After Will be Compared Between the Intervention and Wait-list Control Groups and Within Nursing Homes Before and After the CHATO Training.
Description: NH Level Deidentified Resident data from nursing homes
Time Frame: Baseline, 1 month
Population: Unable to collect information due to lack of available data. Nursing homes in pilot were not in the same chain and data could not be collected at the organizational level.
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Psychotropic Medication Reports for the One-month Period Before Baseline Data Collection and One Month After Will be Compared Between the Intervention and Wait-list Control Groups and Within Nursing Homes Before and After the CHATO Training.
Description: NH Level Deidentified Resident data from nursing homes
Time Frame: Baseline, 1 month
Population: as for outcome 3
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Implementation Strategies Used in Each Nursing Home (Nursing Home Level Data)
Description: The implementation strategies survey is a 35-question descriptive survey developed by the investigators with Advisory Board input, to identify the strategies and approach types used by the NH to implement the training. Eight nursing homes were surveyed. Twenty possible implementation strategies were suggested in the toolkit. The number represents the total strategies used to implement the training in each nursing home.
Time Frame: 1 month (post training)
Population: Eight nursing homes were surveyed. Twenty possible implementation strategies were suggested in the toolkit. The number represents the total strategies used to implement the training in each nursing home.
Measure: Number; unit: Implementation Strategies
Units Other Than Participants: Nursing Homes
Groups:
- Number of Strategies Used to Implement Training: Eight nursing homes were surveyed. Twenty possible implementation strategies were suggested in the toolkit. The number represents the total strategies used to implement the training in each nursing home.
Arm/Group | Number of Strategies Used to Implement Training
Number analyzed (Participants) | 8
Number analyzed (Nursing Homes) | 8
Implementation Strategies
  Feasibility Nursing Home | 7
  Nursing Home 1 | 7
  Nursing Home 2 | 11
  Nursing Home 3 | 3
  Nursing Home 4 | 11
  Nursing Home 5 | 7
  Nursing Home 6 | 9
  Nursing Home 7 | 8

6. Secondary Outcome: Artifacts of Culture Change Scores Per Nursing Home to Assess Nursing Home Practices, Environment, and Staffing (Nursing Home Level Training)
Description: The Artifacts of Culture Change Tool measures NH care environment and practices, leadership and workplace practices, staffing outcomes, and occupancy. Total Artifacts of Culture Change score by nursing home. Scores indicate what percentage of the nursing home environment is person-centered. Range is 0-100%. The average for nursing homes nationwide is 59%
Time Frame: 1 month (post training)
Measure: Number; unit: score on a scale
Units Other Than Participants: Nursing Homes
Groups:
- Artifacts of Culture Change: NH environment and organizational practice was measured using the Artifacts of Culture Change Tool, a 79-item assessment with six subscales: Care Practice, Environment, Family and Community, Leadership, Workplace Practice, and Staffing Outcomes and Occupancy. Responses for each item range from 0 to 5 depending on the scoring for each question and summed for each subscale; the total score is calculated as a sum of the subscales.
Arm/Group | Artifacts of Culture Change
Number analyzed (Participants) | 8
Number analyzed (Nursing Homes) | 8
score on a scale
  Feasibility Nursing Home | 45.3
  Nursing Home 1 | 64.7
  Nursing Home 2 | 66.9
  Nursing Home 3 | 70.2
  Nursing Home 4 | 80.5
  Nursing Home 5 | 36.0
  Nursing Home 6 | 35.2
  Nursing Home 7 | 49.1

7. Secondary Outcome: Nursing Home Implementation Strategies Assessed by Interviews Will be Described, Categorized, and Correlated With Participation Rates.
Description: Leadership Phone Interviews measures qualitative data regarding implementation strategies, lessons learned, and overall evaluation of the CHATO pilot from the NH leadership perspective.
Time Frame: 1 month (post training)
Population: We were unable to conduct interviews with the nursing homes due to the COVID-19 pandemic.
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: The Cost Associated With Hypothesized BPSD Reductions After the CHATO Training Will be Calculated Using Primary Outcomes and Wage Data.
Description: Staff Wage Data measures wages per hour by NH role and will be used in a simple cost-effectiveness analysis (CEA).
Time Frame: 1 month (post training)
Population: We were unable to collect BPSD data from nursing homes.
Arm/Group | Intervention | Waitlist Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline, 1 month, 3 months
Arm/Group | All Direct Care Staff
All-Cause Mortality (participants affected / at risk) | 0/219
Serious Adverse Events (participants affected / at risk) | 0/219
Other Adverse Events (participants affected / at risk) | 0/219

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT03849937/Prot_SAP_000.pdf
  • Informed Consent Form (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT03849937/ICF_001.pdf